CLINICAL TRIAL: NCT06490640
Title: Factors Influencing the Mortality of Patients With Subarachnoid Haemorrhage in the Intensive Care Unit
Brief Title: Factors Influencing the Mortality of Patients With Subarachnoid Haemorrhage
Status: Completed | Type: Observational
Sponsor: Melike Cengiz (Other)
Responsible Party: Sponsor-Investigator, Melike Cengiz, MD,Professor Doctor, Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: Akdeniz U.
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Spontaneous Subarachnoid Hemorrhage
Keywords: Intensive Care Unit; Mortality; Spontaneous subarachnoid haemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spontaneous subarachnoid haemorrhage survival cohort: Demographic and clinical data derived and analyzed included age, sex, smoking history, comorbidities. Presenting signs and symptoms, diagnoses responsible for spontaneous SAH (aneurysm, arterial malformation, etc.), site of aneurysm, risk factors, location of the aneurysm, risk factors, blood pressure during ICU admission, and scores from grading systems indicating clinical and radiological severity of the disease were recorded. Procedures for spontaneous SAH, complications during ICU follow-up (vasospasm, meningitis, electrolyte disturbances, rebleeding, DCI, VIP, sepsis/septic shock) and treatments, duration of ICU stay and mechanical ventilation, ICU outcome (survival or mortality), causes of mortality and brain death status were recorded.
  Interventions: Other: Spontaneous subarachnoid haemorrhage survival cohort
- Spontaneous subarachnoid haemorrhage mortality cohort: Demographic and clinical data derived and analyzed included age, sex, smoking history, comorbidities. Presenting signs and symptoms, diagnoses responsible for spontaneous SAH (aneurysm, arterial malformation, etc.), site of aneurysm, risk factors, location of the aneurysm, risk factors, blood pressure during ICU admission, and scores from grading systems indicating clinical and radiological severity of the disease were recorded. Procedures for spontaneous SAH, complications during ICU follow-up (vasospasm, meningitis, electrolyte disturbances, rebleeding, DCI, VIP, sepsis/septic shock) and treatments, duration of ICU stay and mechanical ventilation, ICU outcome (survival or mortality), causes of mortality and brain death status were recorded.
  Interventions: Other: Spontaneous subarachnoid haemorrhage mortality cohort

INTERVENTIONS:
Other: Spontaneous subarachnoid haemorrhage survival cohort — consists of surviving patients
  Groups: Spontaneous subarachnoid haemorrhage survival cohort
Other: Spontaneous subarachnoid haemorrhage mortality cohort — consists of deceased patients
  Groups: Spontaneous subarachnoid haemorrhage mortality cohort

SUMMARY:
Spontaneous subarachnoid haemorrhage (SAH) is a serious cerebrovascular disease with high morbidity and mortality.Determining the factors associated with mortality in the ICU follow-up and treatment of patients with spontaneous SAH is very important for clarifying these uncertainties and improving ICU outcomes.In the literature, there are very few studies analysing ICU mortality and mortality-related factors in this patient group.The aim of this study was to determine the demographic/clinical characteristics and factors affecting the mortality of spontaneous SAH patients admitted in the ICU.

DETAILED DESCRIPTION:
Patients aged 18 years and older who were diagnosis of spontaneous SAH and admitted the ICU were included in the study. The diagnosis of spontaneous SAH was based on the brain computed tomography (CT) or lumbar puncture. Patients with a final outcome (survival or mortality) in our centre were included in the analysis were included. Only patients admitted to the ICU for the first time were included. Patients with traumatic SAH, history of significant head trauma in the previous two weeks (any abnormality on brain CT requiring hospitalisation for more than 24 hours), pregnancy and length of ICU stay ≤24 hours were excluded.The clinical and radiological severity of the patients at ICU admission was according to Acute Physiological and Chronic Health Evaluation-II score (APACHE II), Glasgow Coma Scale (GCS), Modified Fisher Scale, World Federation of Neurological Societies (WFNS) and Hunt and Hess (H&H) grading systems.Demographic and clinical data derived and analyzed included age, sex, smoking history, comorbidities. Presenting signs and symptoms, diagnoses responsible for spontaneous SAH (aneurysm, arterial malformation, etc.), site of aneurysm, risk factors, location of the aneurysm, risk factors, blood pressure during ICU admission, and scores from grading systems indicating clinical and radiological severity of the disease were recorded. Procedures for spontaneous SAH, complications during ICU follow-up (vasospasm, meningitis, electrolyte disturbances, rebleeding, DCI, VIP, sepsis/septic shock) and treatments, duration of ICU stay and mechanical ventilation, ICU outcome (survival or mortality), causes of mortality and brain death status were recorded. According to the outcome of the ICU process, the patients were divided into two groups as survival and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with a confrmed diagnosis of spontaneous subarachnoid haemorrhage by a brain computed tomography (CT)
* Patients with a final outcome (survival or mortality) in our centre

Exclusion Criteria:

* Patients with traumatic SAH
* History of significant head trauma in the previous two weeks (any abnormality on brain CT requiring hospitalisation for more than 24 hours)
* Pregnancy
* Length of intensive care unit stay ≤24 hours

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who were diagnosis of spontaneous SAH and admitted the intensive care unit were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
determine mortality and causes | 01 January 2019-31 December 2023
  determine mortality and its causes in patients with spontaneous subarachnoid haemorrhage

SECONDARY OUTCOMES:
factors affecting mortality | 01 January 2019-31 December 2023
  evaluate the clinical characteristics and factors affecting mortality in subarachnoid haemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Arslan Yildiz, MD, Principal Investigator — Akdeniz University School of Medicine, Department of Anesthesiology and Intensive Care, Turkey; Murat Yilmaz, Professor, Principal Investigator — Akdeniz University School of Medicine, Department of Anesthesiology and Intensive Care, Turkey; Onur Cetinkaya, MD, Principal Investigator — Akdeniz University School of Medicine, Department of Anesthesiology and Intensive Care, Turkey
Locations (1):
- Akdeniz University School of Medicine, Department of Anesthesiology and Intensive Care, Turkey, Antalya, Turkey (Türkiye)